CLINICAL TRIAL: NCT04331301
Title: Bipolar Needlescopic Enucleation Versus Vapoenucleation of the Prostate: A Prospective Randomized Study
Brief Title: Bipolar Needlescopic Enucleation Versus Vapoenucleation of BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDIRB2017122601-09
Record Dates: First submitted 2020-03-29; First posted 2020-04-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Prostate Obstruction; Prostatic Hyperplasia; Prostatic Hypertrophy, Benign
Keywords: BPH, IPSS, Bipolar
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: interventions are blinded to both patients and doctors who 1ry assess and follow-up patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vapoenucleation group (Active Comparator): Group A
  Interventions: Procedure: Bipolar Vapo-Enucleation of the prostate
- needlescopic enucleation (Active Comparator): group B
  Interventions: Procedure: Bipolar Needlescopic Enucleation of the prostate

INTERVENTIONS:
Procedure: Bipolar Vapo-Enucleation of the prostate — group A: Patient will be subjected to bipolar endoscopic enucleation of the prostate by vaporization electrode (vapoenucleation).
  Other Names: BVEP
  Arms: vapoenucleation group
Procedure: Bipolar Needlescopic Enucleation of the prostate — group B: Patient will be subjected to bipolar endoscopic enucleation of the prostate by hot knife electrode (Needlescopic Enucleation ).
  Other Names: BNEP
  Arms: needlescopic enucleation

SUMMARY:
Transurethral resection of the prostate (TURP) is the current standard procedure for men with prostate volume 30-80 gm. In case with large prostate adenoma (>80 g), the resection time required by TURP is associated with increased risk of TUR syndrome, blood loss and other complications.

Many types of minimally invasive surgery exist along with new equipment and techniques. Many types of laser devices such as greenlight laser, thulium laser and holmium laser, are used to enucleate the prostate. Increasing evidence has proven their safety and efficacy However, the use of laser devices is difficult and associated with steep learning curve and high medical expenses.

PKEP is a safe and effective procedure for the treatment of bladder obstruction secondary to BPH. This procedure not only improves maximum flow rate at 3 and 12 months after surgery, but it also improves all other recorded parameters (IPSS, QOL, IEFF-5, PVR, PSA).

A button electrode can be effectively used to enucleate the prostate because of its powerful vaporisation and strong coagulation (B-TUEP technique) ,such as that with a holmium laser, thulium laser and greenlight laser. However its associated with short term complication as early irritative symptoms, Bulai reported that 16.7% of the patients suffering from early irritative symptoms while Geavlete reported that 11.4% of patient suffering from early irritative symptoms.

DETAILED DESCRIPTION:
Aim: compare safety and efficacy and adverse events of endoscopic enucleation of large prostate using hot knife electrode (needloscopic enucleation) versus the standard vaporization electrode ( vapoenucleation) patients & methods: Patients will randomly be divided into two equal groups: Group A: Patient will be subjected to bipolar endoscopic enucleation of the prostate by vaporization electrode (vapoenucleation).

Group B: Patient will be subjected to endoscopic enucleation of the prostate by bipolar hot kife electrode (needloscopic enucleation) Inclusion criteria: patients with Qmax of less than 15 mL/second due to BPH, severe LUTS/BPH requiring surgical treatment, and International Prostate Symptom Score (IPSS)>7 due to BPH.

exclusion criteria: prostate and/or bladder cancer, bladder diverticula, urethral stricture, active urinary tract infection (UTI), unless treated, and men with neurogenic voiding dysfunction.

Operative Technique: Endoscopic enucleation of the prostate in saline utilizing either bipolar vaporization electrode or bipolar hot knife (collin's) electrode.

follow up: operative time, resected tissue weight, cath time, hospital stay and change of; IPSS,QOL, Qmax, PVR, PSA, IIEF-5 & MSHQ-EjD besides; perioperative adverse events are recorded & followed-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with Qmax of less than 15 mL/second due to BPH, severe LUTS/BPH requiring surgical treatment, and International Prostate Symptom Score (IPSS)>7 due to BPH.

Exclusion Criteria:

* prostate and/or bladder cancer, bladder diverticula, urethral stricture, active urinary tract infection (UTI), unless treated, and men with neurogenic voiding dysfunction.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 214 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
IPSS | change of IPSS from Basline at 1,3 and 6 months postoperatively
  international prostate symptoms score (range 0 -35, the lower value is better)

SECONDARY OUTCOMES:
QOL | Change of QOL from Basline at 1,3 and 6 months postoperatively
  Quality of life questionnaire (range 0 - 6, the lower value is better)
Qmax | Change of Qmax from Basline at 1,3 and 6 months postoperatively
  maximum urinary flow rate (it ranges from 0(retention) to 25 mL/s or more the higher value is better)
PVRU | Change of PVRU from Basline at 1,3 and 6 months postoperatively
  Post-operative residual urine (volume it ranges from 0 ml (normal) to more than 1 liter the lower value is better
TRUS measured prostate volume | Change of PV from Basline at 1,3 and 6 months postoperatively
  Prostate volume measured by Transrectal Ultrasonography the lower value is better

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Shaer, Principal Investigator — waleed_elshaer@hotmail.com
Locations (1):
- Banha University Hospitals, Banhā, Kalubyia, Egypt